CLINICAL TRIAL: NCT01959750
Title: Psychological Intervention on Burnout in ICU Caregivers: a Randomised Controlled Study
Brief Title: Psychological Intervention on Burnout in ICU Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pr. Bara RICOU, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CER 08-220 (NAC08-069)
Record Dates: First submitted 2013-09-23; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Burnout; Anxiety; Depression
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: problem-based sessions
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: problem-based sessions — weekly sessions for small groups of caregivers, led by two psychologists acting as moderators and using a systemic approach, as suggested in other peer-support groups using a problem-based method
  Arms: Intervention Group

SUMMARY:
ICU caregivers face up to a demanding job with a high level of technical skills, a stressful environment, and a heavy work load. They run a high risk of developing burnout that can impact on their welfare, performance, and patient care. Burnout favours absenteeism and staff quitting their jobs, whereas the shortage of ICU caregivers already started. No randomised controlled intervention aimed at reducing such distresses had been run until now.

This study allowed finding a new method of psychological support applicable in the special environment of ICU. Our findings suggest that psychologists specifically assigned to treat ICU caregivers might be beneficial on their burnout.

ELIGIBILITY:
Inclusion Criteria:

* all ICU caregivers rrom the University Hospital of Geneva

Exclusion Criteria:

* refusals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Measurement of the changes in the levels of anxiety, depression, and burnout in nurses and nursing auxiliaries. | At the beginning , at the end and 6 months after the end of the intervention.
  Anxiety (HA) and depression (HD) were identified by the validated French version of the Hospital Anxiety and Depression Scale (HADS), which is composed of 14 items, self-rated using a 4-point Likert scale (0 to 3). The sub-scale scores of anxiety and depression range respectively from 0 to 7 (no distress), 8 to 10 (borderline), 11 to 15 (significant) and 16 to 21 (severe distress).
  Burnout was evaluated using the Maslach Burnout Inventory (MBI) in its Fontaine French version; it is composed of 22 questions on a 7-point Likert scale (0 to 6). This tool measures the 3 dimensions of burnout independently: emotional exhaustion, depersonalisation, and personal accomplishment. Scores of ≥ 27, ≥ 10, or ≤33 respectively for the 3 dimensions, can be a sign of burnout. A severe burnout can also be defined as the cumulated score of MBI of > -9.

SECONDARY OUTCOMES:
Composite measurement of the changes of ICU activity and absenteeism before, during, just after and six months after the intervention. | 4 three-months time periods (cf. Description).
  ICU activities and absenteeism were analysed during 4 three-month time periods, i.e. 3 months before [Before] (January to March 2009), 3 months during [During] (randomly picked out as September and November 2009, and January 2010), 3 months following the end of the intervention [After] (April to June 2010) and from 7 to 10 months after intervention [At 6 months] (November, December 2010 and January 2011). Absenteeism was defined as the number of caregivers absent at least once per time period, independently of the duration of the absence.

OTHER OUTCOMES:
Measurement of staff quitting their jobs | At the end of the intervention
  We identified how many persons had quitted the ICU between the beginning and the end of the intervention (inclusion time).

CONTACTS AND LOCATIONS:
Overall Officials: Bara Ricou, Professor, Study Director — University Hospitals of Geneva
Locations (1):
- University Hopitals of Geneva, Geneva, Switzerland